CLINICAL TRIAL: NCT04727138
Title: 3-part Study to Assess Safety, Tolerability, PK and PD of Single and Multiple Ascending Doses of EXS21546, and to Evaluate the Relative Bioavailability of 2 Formulations, in Healthy Male Subjects
Brief Title: 3-part Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of EXS21546
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exscientia AI Limited (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EXS21546-001
Record Dates: First submitted 2020-12-23; First posted 2021-01-27 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms | interventions — Suspensions; Capsules; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 and Part 2 are double blind. Part 3 is open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EXS21546 Powder for Oral Suspension (Experimental): EXS21546 Powder for Oral Suspension
  Interventions: Drug: EXS21546 Powder for Oral Suspension; Other: Midazolam; Other: Food Effect
- Placebo (Placebo Comparator): Placebo Powder for Oral Suspension
  Interventions: Other: Midazolam; Other: Food Effect; Other: Placebo Powder for Oral Suspension
- EXS21546 Granule in Capsule (Experimental): EXS21546 Granule in Capsule
  Interventions: Drug: EXS21546 Granule in Capsule; Other: Food Effect

INTERVENTIONS:
Drug: EXS21546 Powder for Oral Suspension — EXS21546 Powder for Oral Suspension
  Arms: EXS21546 Powder for Oral Suspension
Drug: EXS21546 Granule in Capsule — EXS21546 Granule in Capsule
  Arms: EXS21546 Granule in Capsule
Other: Midazolam — Interaction
  Arms: EXS21546 Powder for Oral Suspension; Placebo
Other: Food Effect — Fed/Fasted
Other: Placebo Powder for Oral Suspension — Placebo Powder for Oral Suspension
  Arms: Placebo

SUMMARY:
A 3-part Study to Assess Safety, Tolerability, PK and PD of Single (Part 1) and Multiple (Part 2) Ascending Doses of EXS21546, and to Evaluate the Relative Bioavailability of a Solid Dose Formulation Compared to a Powder for Oral Suspension (Part 3), in Healthy Male Subjects.

DETAILED DESCRIPTION:
Part 1 is a randomised, double-blind, placebo-controlled, SAD study with a food effect assessment.

Part 2 is a randomised, double-blind, placebo controlled, MAD study over 14 days. In order to explore the potential CYP3A4 inducer effect, midazolam will also be administered in one cohort.

Part 3 is a 3-period, open label, randomised, sequential study. Each subject will receive solid dose formulation and powder for oral suspension in a randomised manner.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.0 to 30.0 kg/m2
* Weight ≥60 kg
* Must adhere to contraception requirements

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the 90 days prior to Day 1
* Subjects who have previously been administered IMP in this study.
* Evidence of current SARS-CoV-2 infection
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in males >21 units per week
* A confirmed positive alcohol breath test at screening or admission
* Current smokers and those who have smoked within the last 12 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
* Subjects with pregnant or lactating partners
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results
* Regimen L only: History of sleep apnea
* Subjects with a history of cholecystectomy or gall stones
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
* Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever is allowed unless it is active
* Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-04-16 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent Adverse Events | 1 month
  Number of participants with treatment emergent Adverse Events
EXS21546 and Metabolite Area under the plasma concentration versus time curve (AUC) | 17 days
  EXS21546 and Metabolite Area under the plasma concentration versus time curve (AUC)
EXS21546 and Metabolite Peak Plasma Concentration (Cmax) | 17 days
  EXS21546 and Metabolite Peak Plasma Concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Evans, Principal Investigator — Quotient Sciences Principal Investigator
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No